CLINICAL TRIAL: NCT03751137
Title: Longitudinal, Prospective Comparison of the Gastrointestinal Tract of Breastfed and Formula Fed Infants Via Fecal Analysis of the Microbiome, Intestinal Epithelial Cell Expression of Gut Hormones, and Fecal Analysis of the Metabolome
Brief Title: GI Tract Biomarkers in Infants With Different Diets
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Principal Investigator, Matthew Di Guglielmo, Chief, Division of General Academic Pediatrics, Nemours Children's Clinic
Other Study IDs: 822736
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Obesity, Childhood
Keywords: Microbiome; Gut-brain axis; Satiety; Hormone; Obesity; Metabolome
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fecal samples containing microbial genetic material and, to a lesser degree, human intestinal epithelial cells with human genetic material.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Breast Feeding: Infants who, when enrolled, are exclusively breast feeding.
- Formula Feeding: Infants who, when enrolled, are exclusively formula feeding.

SUMMARY:
Childhood obesity is increasing with more than one-third of adolescents currently overweight and one in five with obesity. The lifelong incidence of obesity-related morbidities is also increasing with childhood obesity. It is not yet known how obesity develops in an individual, specifically in early childhood. Further, it is unclear what mechanistic role a child's earliest nutrition or changing intestinal flora has in the etiology of obesity. Very young children are developing appetite and satiety patterns early in life. Nutrition and gut microbial flora have impact on how these processes unfold, but specific mechanisms are not yet well understood. The investigators hypothesize that formula-fed infants with changes in their microbial flora are more likely to have altered carbohydrate metabolism, evidenced by greater imbalances of fatty acid production, and are more likely to have accelerated growth trajectory due to satiety disruption. The investigators further hypothesize that altered carbohydrate metabolism, e.g. imbalances of short- and long-chain fatty acid levels in the gut, stimulate cellular stress and affect specific gut hormones. This study will compare the microbiome of the intestinal microbial flora in two groups of infants, one breast fed and the other formula fed, using longitudinally collected fecal samples from both groups. Samples will be subjected to shotgun metagenomic analysis and simultaneous metabolomic analysis. A bioinformatics approach will elucidate key differences among and between sample groups, and will further analyze bacterial gene expression levels related to carbohydrate metabolism. This study will compare the expression of human proteins involved in cellular stress response and gut peptide signaling by applying quantitative Reverse Transcriptase-Polymerase Chain Reaction to human messenger RNA isolated from the longitudinally collected samples from both groups. Finally, this study will monitor the trajectory of growth and feeding over the first 2 years of life. The project's focus on the influence of different early feeding types, microbial flora changes, and altered carbohydrate metabolism leading to disruption of gut-brain signaling will provide critical data for host:microbiome interactions and translational therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy, male or female term infants
* Exclusively breast or formula feeding
* Never been exposed to oral or intravenous antibiotics or probiotics

Exclusion Criteria:

* Maternal antibiotic use while breast-feeding
* Infant or maternal use of probiotics
* Current or recent (<14 days) gastrointestinal infection (viral, bacterial, or fungal)
* Gastrointestinal mucosal disease, or significant constipation
* Consuming formula that is not standard cow's milk formula
* Infants on acid suppression medications or infants receiving high-density formula (>20 calories/ounce) may be enrolled and will be analyzed separately

Ages: 6 Weeks to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants who are either exclusively breast feeding or exclusively formula feeding are eligible to enroll if meeting other criteria.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Microbiome | Enrollment
  Metagenomic analysis of microbial organisms in infant's feces
Microbiome | 6 months
  Metagenomic analysis of microbial organisms in infant's feces
Microbiome | 12 months
  Metagenomic analysis of microbial organisms in infant's feces
Microbiome | 18 months
  Metagenomic analysis of microbial organisms in infant's feces

SECONDARY OUTCOMES:
Metabolome | Enrollment
  Metabolic products present in infant's feces
Metabolome | 6 months
  Metabolic products present in infant's feces
Metabolome | 12 months
  Metabolic products present in infant's feces
Metabolome | 18 months
  Metabolic products present in infant's feces
Gut hormone gene expression | Enrollment
  Transcriptional output of human epithelial cells in infant's feces
Gut hormone gene expression | 6 months
  Transcriptional output of human epithelial cells in infant's feces
Gut hormone gene expression | 12 months
  Transcriptional output of human epithelial cells in infant's feces
Gut hormone gene expression | 18 months
  Transcriptional output of human epithelial cells in infant's feces

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Di Guglielmo, MD PhD, Principal Investigator — Nemours
Locations (1):
- Nemours Children's Hospital - Delaware, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
We will release deidentified metagenomic sequencing data from each participant to either database of Genotypes and Phenotypes (dbGaP) or Sequence Read Archive (SRA).
Supporting Information: SAP, Analytic Code
Time Frame: At the conclusion of the study
Access Criteria: To be determined

REFERENCES:
- [Background] Di Guglielmo MD, Franke KR, Robbins A, Crowgey EL. Impact of Early Feeding: Metagenomics Analysis of the Infant Gut Microbiome. Front Cell Infect Microbiol. 2022 Mar 4;12:816601. doi: 10.3389/fcimb.2022.816601. eCollection 2022. PMID 35310842
- [Background] Di Guglielmo MD, Franke K, Cox C, Crowgey EL. Whole genome metagenomic analysis of the gut microbiome of differently fed infants identifies differences in microbial composition and functional genes, including an absent CRISPR/Cas9 gene in the formula-fed cohort. Hum Microb J. 2019 Jun;12:100057. doi: 10.1016/j.humic.2019.100057. Epub 2019 May 25. PMID 34278055